CLINICAL TRIAL: NCT01783535
Title: Protocol for the Study and Treatment of Participants With Intraocular Retinoblastoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SJRET6; NCI-2013-00409 (Registry Identifier: NCI Clinical Trials Reporting Program)
Record Dates: First submitted 2013-01-31; First posted 2013-02-05 (Estimated); Last update posted 2024-04-16 (Actual); Status verified 2024-03

CONDITIONS: Retinoblastoma
Keywords: intraocular retinoblastoma
MeSH Terms: conditions — Retinoblastoma | interventions — Vincristine; Topotecan; trioctyl phosphine oxide; Filgrastim; Granulocyte Colony-Stimulating Factor; pegfilgrastim; Carboplatin; Cryotherapy; Brachytherapy; Etoposide; Cyclophosphamide; Mesna; Doxorubicin; Eye Enucleation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Stratum A (Experimental): Participants with early bilateral or unilateral (unifocal or multifocal) retinoblastoma (R-E I-III, IC A-B; R-E IV with IC A or B; or IC C with limited sub-retinal seeding), and participants with bilateral disease in whom the advanced eye has been enucleated upfront (without any high risk histopathology) and the remaining eye has early stage disease (as defined above).
  Interventions (see detailed description): vincristine, carboplatin, topotecan, filgrastim or PEG-filgrastim, and focal therapy, including cryotherapy, laser photocoagulation, thermo-therapy, plaque radiotherapy.
  Interventions: Drug: vincristine; Drug: topotecan; Drug: filgrastim; Drug: PEG-filgrastim; Drug: carboplatin; Other: focal therapy
- Stratum B (Experimental): Participants considered candidates for conservative management including those:
  1. Participants with bilateral retinoblastoma who have R-E IV-V and IC D in one eye
  2. Participants with advanced unilateral (unifocal or multifocal) retinoblastoma (R-E IV-V and IC D-E) who demonstrate foveal sparing by the tumor during EUA. Due to foveal sparing, these patients have potential for vision preservation.
  Interventions (see Detailed Description): vincristine, topotecan, carboplatin, etoposide, filgrastim or PEG-filgrastim and focal therapy, including cryotherapy, laser photocoagulation, thermo-therapy, plaque radiotherapy.
  Interventions: Drug: vincristine; Drug: topotecan; Drug: filgrastim; Drug: PEG-filgrastim; Drug: carboplatin; Other: focal therapy; Drug: etoposide
- Stratum C (Experimental): Participants with advanced (R-E IV-V and IC D-E) unilateral retinoblastoma who require upfront enucleation. Participants will be assessed and treated by low, intermediate or high risk.
  Interventions (see Detailed Description): vincristine, cyclophosphamide, MESNA, doxorubicin, etoposide, carboplatin, filgrastim or PEG-filgrastim, enucleation
  Interventions: Drug: vincristine; Drug: filgrastim; Drug: PEG-filgrastim; Drug: carboplatin; Drug: etoposide; Drug: cyclophosphamide; Drug: MESNA; Drug: doxorubicin; Procedure: enucleation
- Stratum D (Experimental): Participants with bilateral retinoblastoma who may require upfront enucleation for one eye due to advanced disease (R-E IV-V and IC E).
  Interventions (see Detailed Description): vincristine, carboplatin, topotecan, etoposide, enucleation, filgrastim or PEG-filgrastim, focal therapy, including cryotherapy, laser photocoagulation, thermotherapy (and thermo-chemotherapy) and episcleral plaque brachytherapy, and external beam radiation or proton beam radiation in select cases.
  Interventions: Drug: vincristine; Drug: topotecan; Drug: filgrastim; Drug: PEG-filgrastim; Drug: carboplatin; Other: focal therapy; Drug: etoposide; Procedure: enucleation; Radiation: external beam radiation or proton beam radiation

INTERVENTIONS:
Drug: vincristine — Given via minibag/gravity flow.
  Other Names: VCR; Oncovin(R)
Drug: topotecan — Given IV over 30 minutes.
  Other Names: TOPO; Hycamtin(R)
  Arms: Stratum A; Stratum B; Stratum D
Drug: filgrastim — Given subcutaneously 24-36 hours after chemotherapy for 7-10 days, until absolute neutrophil count (ANC) is >2,000/µL on one occasion after the expected nadir.
  Other Names: G-CSF; Neupogen(R)
Drug: PEG-filgrastim — Given subcutaneously 24-36 hours after chemotherapy for 7-10 days, until ANC is >2,000/µL on one occasion after the expected nadir.
  Other Names: pegylated filgrastim; PEG filgrastim; SD-01; Neulasta(R)
Drug: carboplatin — Given IV over 60 minutes. Given periocular (subtenon/subconjunctival).
  Other Names: CARBO; Paraplatin(R)
Other: focal therapy — Focal treatments will be administered at the discretion of the treating team to strata A, B and D. In select cases of very early stage retinoblastoma (Stratum A), participants may receive focal therapies only and chemotherapy will be held at the discretion of the treating team. If there is any evidence of progression or unsatisfactory results, the participant will begin chemotherapy as per Stratum A. For selected participants an effort will be made to perform sequential chemo-thermotherapy. In these cases, carboplatin will be administered one or two hours prior to thermotherapy.
  Other Names: cryotherapy; laser photocoagulation; thermo-therapy; plaque radiotherapy; thermo-chemotherapy; episcleral plaque brachytherapy
  Arms: Stratum A; Stratum B; Stratum D
Drug: etoposide — Given IV. Participants who cannot tolerate etoposide may be given etoposide phosphate (Etopophos(R)).
  Other Names: ETOP; VP-16; Vepesid(R); Etopophos(R)
  Arms: Stratum B; Stratum C; Stratum D
Drug: cyclophosphamide — Given IV.
  Other Names: CYCLO; Cytoxan(R)
  Arms: Stratum C
Drug: MESNA — Given IV before CYCLO and at 3, 6 and 9 hours after CYCLO.
  Other Names: Mesnex(R)
  Arms: Stratum C
Drug: doxorubicin — Given IV on Day 1 of Cycles 2, 4 and 6 in Stratum C high-risk.
  Other Names: DOXO; Adriamycin(R)
  Arms: Stratum C
Procedure: enucleation — Eye removal due to advanced disease in Strata C and D participants.
  Other Names: eye removal
  Arms: Stratum C; Stratum D
Radiation: external beam radiation or proton beam radiation — EBRT or proton beam radiation will be administered to any eye in which the disease is considered to be not controllable with focal treatments alone, and in participants with enucleated eyes in which high risk of orbital and/or central nervous system disease is documented histologically (high-risk group with disease extension beyond the sclera or cornea, or beyond the cut end of the optic nerve). EBRT will be administered using standard techniques practices with the objective of limiting dose to normal tissues including the hypothalamic-pituitary unit, supratentorial brain, orbit, cochleae and contralateral eye when indicated. Participants will be evaluated on an individual basis to determine whether they might benefit from referral for proton therapy.
  Other Names: EBRT
  Arms: Stratum D

SUMMARY:
The primary objective of this protocol is to evaluate the response rate of bilateral disease participants who have at least one eye with advanced intra-ocular retinoblastoma (stratum B) using upfront therapy with chemotherapy delivered directly to the eye. The main biology objective is to improve our understanding of the biology and tumorigenesis (how tumor develops) of retinoblastoma when biology specimens are available. As clinicians, the primary goal of the investigators for children with retinoblastoma is to provide optimal therapy using multiple treatment approaches [chemotherapy (into the vein and directly into membrane of eyeball), cryotherapy (freeze and destroy tumor), thermotherapy (laser or heat to destroy tumor), radiation therapy, and surgical removal of eye if needed) in an attempt to preserve the eye and vision whenever possible, while still curing the disease. Therefore, all children with non-metastatic retinoblastoma at St. Jude will be offered enrollment on this study.

PRIMARY OBJECTIVE:

* To evaluate the response (complete + partial response) rate of bilateral disease participants who have at least one eye with advanced intraocular retinoblastoma (Stratum B) to two upfront courses of therapy consisting of subconjunctival carboplatin and systemic topotecan.

SECONDARY OBJECTIVES:

* To evaluate the ocular survival of eyes and event-free survival of participants by strata.
* To prospectively analyze intraocular disease tissue for participants with at least one eye undergoing enucleation in order to identify the mechanism of RB1 bi-allelic inactivation. Participants may undergo upfront enucleation (due to advanced disease at diagnosis) or may receive enucleation due to progressive disease during protocol therapy.

DETAILED DESCRIPTION:
Participants will be stratified into four main treatment groups, depending on whether retinoblastoma is present in one or both eyes and disease grouping [early or advanced, Reese-Ellsworth (R-E) group I-V, and International Classification A-E]. Additionally, participants will be invited to participate in exploratory research objectives that address cognitive and functional development of children with retinoblastoma, the pharmacokinetics of topotecan in young children, and evaluation of ototoxicity, including genetic analysis.

TREATMENT PLAN

STRATUM A:

* Children ≥ or equal to 6 months old at time of enrollment - 8 courses of vincristine and carboplatin, given at 3-4 week intervals.
* Infants < 6 months old at time of enrollment - Therapy will consist of six courses of chemotherapy; three courses of vincristine and carboplatin, given at 3-4 week intervals, alternating with 3 cycles of vincristine and topotecan, given at 3-4 week intervals.

Focal treatments will be administered at the discretion of the treating team. Focal therapies will include cryotherapy, laser photocoagulation, thermo-therapy and plaque radiotherapy.

STRATUM B:

* Participants without extensive sub-retinal (SR) seeding, treatment will consist of two up-front courses of vincristine and topotecan, given at 3-4 week intervals.
* Participants without SR seeding: ≥ or equal to partial response after 2 cycles, will receive three additional courses of vincristine-topotecan (VT) and six courses of vincristine-carboplatin, given at 3-4 week intervals.
* Participants without SR seeding and < partial response after 2 cycles VT will receive 6 courses of vincristine-carboplatin-etoposide (VCE), given at 3-4 week intervals.
* Participants with extensive sub-retinal (SR) seeding will receive two up-front courses of subconjunctival (also called subtenon or periocular) CARBOplatin and systemic topotecan, given at 3-4 week intervals.
* Participants with SR seeding: > or equal to partial response after 2 cycles will receive three additional courses of vincristine-topotecan, and six courses of vincristine-carboplatin, given at 3-4 week intervals.
* Participants with SR seeding: < partial response after 2 cycles will receive 6 courses of VCE, given at 3-4 week intervals.

Focal treatments will be administered at the discretion of the treating team. Focal therapies will include cryotherapy, laser photocoagulation, thermo-therapy and plaque radiotherapy.

STRATUM C:

Participants with unilateral (unifocal or multifocal) advanced (R-E IV-V and IC D-E) intraocular disease will undergo enucleation. Adjuvant therapy will be based on histopathology:

* low risk participants: Participants in whom the enucleated eye does not show extra-retinal disease (see definition of intermediate and high risk below); will not receive any additional treatment.
* intermediate risk participants: Participants in whom the enucleated eye shows presence of tumor in the anterior chamber, invasion of the ciliary body/iris, massive invasion of the choroid, and invasion of the optic nerve beyond the lamina cribrosa with concomitant invasion of the choroid, will receive 4 courses of adjuvant chemotherapy with vincristine-carboplatin-doxorubicin (VCD).
* high risk participants: Participants in whom the enucleated eye shows involvement of the sclera, or involvement of the optic nerve at the level of the cut-end, will be treated with 6 courses of chemotherapy, with alternating courses of VCE and VCD.
* High-risk participants with extra-ocular extension (i.e. tumor extending beyond the sclera/cornea or beyond the cut end of the optic nerve) will be candidates for external-beam radiation therapy (EBRT) to the entire orbit, including the optic nerve, administered after 2 or 3 courses of treatment. Patients with extra-ocular extension may be considered for enrollment on an alternative therapeutic protocol for metastatic retinoblastoma (or best clinical management).

STRATUM D:

Management of participants with bilateral retinoblastoma is often complex; and some participants will have one eye enucleated upfront due to advanced disease. The decision for enucleation will be made after thorough consideration by the treating team. The treatment of the remaining eye will depend on a combination of two factors: a) R-E group of the remaining eye, and b) Histology of the enucleated eye. Though we have accumulated some information regarding the use of vincristine, cyclophosphamide, and doxorubicin in the treatment of intraocular retinoblastoma, it is not considered standard of care. Therefore, participants with intermediate and high risk features will be treated with 6 courses of vincristine, carboplatin, and etoposide (VCE). Those participants in whom the enucleated eye shows only low risk histology will be eligible to proceed with either stratum A or stratum B therapy. For those receiving stratum B therapy, consideration of periocular carboplatin will be allowed. External beam or proton beam radiation therapy will be considered for patients with extra-ocular extension.

Focal treatments will be administered at the discretion of the treating team. Focal therapies will include cryotherapy, laser photocoagulation, thermo-therapy and plaque radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, untreated intraocular retinoblastoma. Participants previously diagnosed with unilateral retinoblastoma treated surgically, with focal therapy or needing chemotherapy who develop asynchronous involvement of the contralateral eye, or patients with unilateral retinoblastoma treated only with enucleation or focal therapy who develop asynchronous involvement of the contralateral eye, will be eligible for study.
* ECOG Performance Score must be ≤ 2 within two weeks prior to registration.
* Participants must have an adequate liver function, as defined by bilirubin ≤ to 3X upper limit of normal (ULN), and SGOT and SGPT ≤ to 3X ULN.
* Participants must have adequate renal function as defined by serum creatinine ≤ to 3X ULN for age.
* Legal guardians must sign an informed consent indicating that they are aware of this study, the possible benefits, and toxic side effects. Legal guardians will be given a signed copy of the consent form.

Exclusion Criteria:

* Previously treated participants.
* Presence of metastatic disease or gross (residual) orbital involvement
* Participants must not have an invasive infection at time of protocol entry.
* Inability or unwillingness of research participant or legal guardian/representative to give written informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2013-06-19 (Actual); Primary Completion 2023-03-17 (Actual); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Response rate (complete or partial response) | After two upfront courses of chemotherapy (approximately two months after patient enrollment)
  Stratum B patients, those Stratum B patients who had no significant subretinal seeding and received vincristine and topotecan are not evaluable for this primary objective.

SECONDARY OUTCOMES:
ocular survival | at end of study (approximately three years after the last patient enrollment)
  Ocular survival per eye will be defined as the time interval from study enrollment to date of enucleation or to date of last contact for eyes that have not been enucleated.
Event-free survival | at end of study (approximately three years after the last patient enrollment)
  Event-free survival per eye will be defined as the time interval from date on study to date of first event (where an event includes external beam radiation or enucleation) or to the date of last contact for eyes without events.
The mechanism (or frequencies) for each RB1 biallelic inactivation | At end of study (approximately one year after the last patient is enrolled on study)
  The tumor tissue samples will be obtained from participant who has at least one eye undergoing enucleation.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Rodriguez-Galindo, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols